CLINICAL TRIAL: NCT06555224
Title: Role of Postoperative Lubrication in Preventing Dry Eye After Cataract Surgery
Brief Title: Role of Postoperative Lubrication in Cataract Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vienna Institute for Research in Ocular Surgery (Other)
Responsible Party: Principal Investigator, Prim. Prof. Dr. Oliver Findl, MBA, Prim. Prof. Dr., Vienna Institute for Research in Ocular Surgery
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: EK_21_098_0521
Record Dates: First submitted 2024-08-12; First posted 2024-08-15 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigator will be masked to study group allocation
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High Risk Standard of Care (No Intervention): OSFI >= 0.3, NSAID 2x daily for 4 weeks
- High Risk Treatment Group (Experimental): OSFI >= 0.3, NSAID 2x daily for 4 weeks, Systane Hydration MDPF 4x daily for 3 months
  Interventions: Device: Systane Hydration MDPF eye drops
- Low Risk, Reference Group (No Intervention): OSFI < 0.3, NSAID 2x daily for 4 weeks

INTERVENTIONS:
Device: Systane Hydration MDPF eye drops — Systane Hydration MDPF eye drops 4x daily for 3 months additional to routine medication after cataract surgery
  Arms: High Risk Treatment Group

SUMMARY:
Cataract and dry eye are two conditions occurring frequently in the elderly. Several reports suggested a deterioration of dry eye after cataract surgery, causing a significant impact on patients' postoperative satisfaction as well as quality of life. Recently, a novel index, assessing the risk of developing dry eye after cataract surgery in a non-dry eye population, was published; the so called - Ocular Surface Frailty Index (OSFI). This score utilizes 10 items including clinical ocular findings, medical history as well as environmental factors and grade the respective subject in low-risk- or high-risk group. Using the cutoff of 0.3, the rate of postoperative dry eye was 9,6% in the low-risk group and 50% in the high-risk group (p<0.001).

Systane Hydration MDPF eye drops (Alcon Research, Ltd., Fort, Worth, Texas, USA, a division of Novartis) is an artificial tear substitute based on the dual-polymer formula containing HP-Guar and hyaluronic acid. Previous studies found an increase in tear film stability and reduction of subjective complaints. In an animal model corneas treated with Systane Hydration showed the fastest re-epithelialization compared to other HA products supporting the beneficial role of HA-containing artificial tears in corneal wound healing.

The current study seeks to investigate if intensive lubrication, using Systane Hydration MDPF, in the postoperative phase of cataract surgery can reduce the rate of dry eye in the high-risk group. The findings will have a great impact how to identify these patients, to administer the adequate therapy, which might hinder development of dry eye related to cataract surgery.

The goal of this clinical trial is to learn if Systane Hydration MDPF eye drops (Alcon Research, Ltd., Fort, Worth, Texas, USA, a division of Novartis) works to treat prevent postoperative dry eye in adults undergoing cataract surgery. The main questions it aims to answer are:

- to investigate if intensive lubrication, using Systane Hydration MDPF, in the postoperative phase of cataract surgery can reduce the rate of dry eye in a high-risk group. The findings will have a great impact how to identify these patients, to administer the adequate therapy, which might hinder development of dry eye related to cataract surgery.

Participants will:

Take Systane Hydration MDPF eye drops 4x daily for 3 months additional to or just the standard of care medication (NSAID topical 2x daily for 4 weeks) after surgery Visit the clinic after 7 days, 1 month and 3 months after cataract surgery

ELIGIBILITY:
Inclusion Criteria:

* Age older than 18 years
* Cataract surgery scheduled in one or both eyes
* Scheduled for monofocal or monofocal-toric IOL implantation
* OSDI lower than 14
* OSFI higher or equal to 0.3 - Group 1 and Group 2
* OSFI lower than 0.3 - Group 3

Exclusion Criteria:

* Presence of dry eye symptoms preoperatively
* Occurrence of complications during surgery
* Usage of systemic antibiotic therapy
* Any pathology of the ocular surface except dry eye disease (e.g. corneal scarring, cornea ectasia)
* Ocular surgery within prior 3 months
* Ocular injury within prior 3 months
* Ocular herpes of eye or eyelid within prior 3 months
* Active ocular infection
* Active ocular inflammation or history of chronic, recurrent ocular inflammation within prior 3 months
* Eyelid abnormalities that affect lid function
* Ocular surface abnormality that may compromise corneal integrity
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-06-22 (Actual); Primary Completion 2023-12-18 (Actual); Study Completion 2023-12-18 (Actual)

PRIMARY OUTCOMES:
Rate of dry eye symptoms defined by OSDI score >= 13 at 3 months visit | 3 months visit

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Findl, MD, Principal Investigator — Vienna Institute for Research in Ocular Surgery
Locations (1):
- Hanusch Hospital, Department of Ophthalmology, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No
IPD will be availabe upon reasonable request.

REFERENCES:
- [Derived] Palkovits S, Schlatter A, Ruiss M, Fisus A, Bayer N, Kofler P, Findl O. Role of postoperative lubrication in preventing dry eye after cataract surgery in high- and low-risk patients stratified by ocular surface frailty index. PLoS One. 2025 Mar 26;20(3):e0312712. doi: 10.1371/journal.pone.0312712. eCollection 2025. PMID 40138387